CLINICAL TRIAL: NCT03496935
Title: A Randomized Controlled Trial of Tunneled Dialysis Catheters Versus Non-tunneled Dialysis Catheters for Renal Replacement Therapy in the ICU
Brief Title: Tunneled Dialysis Catheters Versus Non-tunneled Dialysis Catheters as First-line for Renal Replacement Therapy in the ICU
Acronym: BACKDOOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Yvelynne Kelly M.D. MSc., Nephrology Fellow, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018P000711
Record Dates: First submitted 2018-03-28; First posted 2018-04-12 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Acute Kidney Injury
Keywords: Renal replacement therapy
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tunneled dialysis catheter (Active Comparator): In this arm, patients will be randomized to undergo tunneled dialysis catheter insertion.
  Interventions: Device: Tunneled versus non-tunneled dialysis catheter insertion
- Non-tunneled dialysis catheter (Active Comparator): In this arm, patients will be randomized to undergo non-tunneled dialysis catheter insertion.
  Interventions: Device: Tunneled versus non-tunneled dialysis catheter insertion

INTERVENTIONS:
Device: Tunneled versus non-tunneled dialysis catheter insertion — The study participants will be randomized either to tunneled or non-tunneled dialysis catheter insertion to commence renal replacement therapy for an acute kidney injury requiring either continuous or intermittent dialysis in the ICU.

SUMMARY:
The investigators propose a randomized controlled trial to examine whether tunneled dialysis catheters should be first-line for acute kidney injury requiring renal replacement therapy (AKI-RRT) in the critical care setting, barring any clinical contraindications, compared to non-tunneled access. This randomized controlled trial will include patients admitted to an intensive care unit (ICU) at Brigham and Women's Hospital (BWH). The investigators will randomize all eligible consented incident patients with AKI requiring renal replacement therapy either to tunneled dialysis catheter or non-tunneled dialysis catheter placement. The inclusion criteria encompasses all adult patients in the BWH ICUs with an incident AKI requiring renal replacement therapy. The investigators' hypothesis is that the rate of overall complications is lower with tunneled dialysis catheters compared to non-tunneled catheters.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is defined by an abrupt decrease in kidney function resulting in the retention of urea and other nitrogenous waste products and in the dysregulation of extracellular volume and electrolytes. AKI is common, harmful and potentially treatable.

Despite decades of research, renal replacement therapy (RRT) in the form of dialysis remains the primary therapy to treat AKI and its complications. Due to convenience of scheduling and distribution of expertise, non-tunneled dialysis catheters have generally been the first-line source of vascular access for patients requiring acute dialysis for AKI in the ICU setting. However, there is evidence that tunneled dialysis catheters are associated with improved outcomes compared to non-tunneled dialysis catheters.

The investigators for this proposed trial performed an observational study at Brigham and Women's Hospital in 2016 comparing outcomes from temporary dialysis catheter versus tunneled dialysis catheter use for renal replacement therapy in the ICU.12 They found that there was a significant increase in median venous and arterial access pressure between temporary dialysis catheters and tunneled dialysis catheters for patients on CVVH with an increased rate ratio of interruptions and decreased blood flow rates for temporary dialysis catheters compared to tunneled dialysis catheters

The investigators now propose a prospective randomized controlled trial to examine whether tunneled dialysis catheters should be first-line for AKI-RRT in the critical care setting, barring any clinical contraindications, compared to non-tunneled access. This RCT will include patients admitted to an ICU at Brigham and Women's Hospital. The investigators will randomize all eligible consented incident patients with AKI requiring renal replacement therapy either to tunneled dialysis catheter or non-tunneled dialysis catheter placement. The inclusion criteria encompasses all adult patients in the BWH ICUs with an incident AKI requiring renal replacement therapy. Exclusion criteria will include 1) clinical instability requiring bedside catheter placement; 2) international normalized ratio (INR) >2.0 or other significant coagulopathy; 3) pending blood cultures within 48 hours or active bacteremia; or 4) urgency of line placement warranting placement within 6 hours. To avoid bias introduced by operator performance, the same group of interventional nephrologists will be utilized to place the catheters in both arms of the trial. The investigators' hypothesis is that the rate of overall complications is lower with tunneled dialysis catheters compared to non-tunneled catheters. Other secondary outcomes of interest include dialysis delivery parameters including access pressures and blood flow rates. The investigators also plan to assessing the feasibility of tunneled dialysis catheter placement for AKI, by capturing data on time to placement, resource utilization and cost. The proposal challenges a common clinical practice; placement of non-tunneled catheters for RRT initiation, which is not evidence-based, to determine if tunneled catheters can improve outcomes for patients compared to usual care.

The investigators will identify all patients with AKI requiring vascular access by reviewing inpatient renal consult patient lists and electronic orders for intermittent hemodialysis (IHD) or continuous renal replacement therapy (CRRT) initiation. Data will be prospectively collected on demographics, comorbidities, laboratory data, and microbiology results on a daily basis. Data will also be abstracted from procedure notes to identify procedural complications. Similarly, CVVH and IHD data (blood flow rates, venous and arterial pressures, total time of RRT per session, and number of interruptions during RRT) will be gathered prospectively on a daily basis from RRT flowsheets and RRT nursing notes. Patients will be followed throughout the entirety of the hospitalization until hospital discharge or death.

ELIGIBILITY:
Inclusion Criteria:

All adult patients in the BWH ICUs with an incident AKI requiring renal replacement therapy

Exclusion Criteria:

1. Clinical instability requiring bedside catheter placement
2. INR >2.0 or other significant coagulopathy
3. Pending blood cultures within 48 hours or active bacteremia
4. Urgency of line placement warranting placement within 6 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of complications | Up to 60 days
  Composite outcome including rate of infection and thrombosis. The incidence of both of these adverse events will be added together to give a composite rate of complications.

SECONDARY OUTCOMES:
Dialysis venous access pressure | Up to 60 days
  Median venous access pressure
Dialysis arterial access pressure | Up to 60 days
  Median arterial access pressure
Dialysis blood flow rate | Up to 60 days
  Median blood flow rate
Feasibility of tunneled catheter placement for AKI | Up to 60 days
  Time to catheter placement
Cost of dialysis access placement for AKI | Up to 60 days
  Cost of dialysis catheter placement

CONTACTS AND LOCATIONS:
Overall Officials: Mallika Mendu, M.D. MBA., Principal Investigator — Brigham and Women's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tsujimoto Y, Miki S, Shimada H, Tsujimoto H, Yasuda H, Kataoka Y, Fujii T. Non-pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2021 Sep 14;9(9):CD013330. doi: 10.1002/14651858.CD013330.pub2. PMID 34519356